CLINICAL TRIAL: NCT06684340
Title: Construction of AI-enabled Models for Predicting the Risk of Sepsis After Major Abdominal Surgery: a Retrospective Multicenter Clinical Study
Brief Title: Risk Factors Identification of Sepsis and Septic Shock After Major Abdominal Surgery Based on Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-24-009
Record Dates: First submitted 2024-11-03; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Sepsis; Postoperative Complications
MeSH Terms: conditions — Sepsis; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Exposure to major abdominal surgery — This study is a retrospective cohort study. The 'exposure' situation is based on historical records and observation, and no active intervention has been conducted on the study subjects to change their exposure status.

SUMMARY:
The goal of this observational study is to identify the risk factors and build the early warning system of sepsis and septic shock after major abdominal surgery based on artificial intelligence. The main questions it aims to answer are:

What are the high risk factors of postoperative sepsis? Which factors can accelerate the progression of sepsis? Researchers will collect perioperative characteristics to construct predictive models of postoperative sepsis in a retrospective abdominal surgical population based on artificial intelligence, and the accuracy of the models were tested in an external dataset.

ELIGIBILITY:
Inclusion Criteria：

1. Patients undergoing major abdominal surgery.
2. The surgeon performing the operation has extensive experience in specialized surgeries such as upper gastrointestinal, hepatobiliary and pancreatic, colorectal, gynecological, and urological surgeries, having completed at least 50 corresponding specialized surgical cases.
3. The anesthesiologist performing the operation has more than 5 years of clinical experience.
4. All surgical patients receive general anesthesia.
5. Patients are aged ≥ 18 years. Exclusion Criteria：

1. Pregnancy-related surgeries (cesarean section, abortion surgery). 2. Patients with known preoperative infection or suspected infection. 3. Severely malnourished patients (BMI reference values are 17 kg/m² for patients < 70 years old and 17.8 kg/m² for patients > 70 years old).

4. Patients who have previously undergone abdominal surgery. 5. Patients without sufficient data, including demographic variables (such as age, gender), surgical details (surgery duration, surgical grade, anesthesia grade, anesthesia duration), and hospitalization details (such as ICU stay, in-hospital mortality).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Internal Cohort: Patients who received major abdominal surgery in each participating hospital before June 2024.
  External Cohort: Patients who received major abdominal surgery, received general anesthesia, and were aged 18 years or older from 2008 to 2019. The data was extracted from the MIMIC - IV (Medical Information Mart for Intensive Care, 2.2 version) database.
Sampling Method: Non-Probability Sample
Enrollment: 22646 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Sepsis within 28 days after surgery. | In the 28-day period following surgery
  For patients within 28 days after surgery, if there is a recorded or suspected infection and the Sequential Organ Failure Assessment (SOFA) score is ≥ 2 points, sepsis can be diagnosed. For sepsis patients, if they still have persistent hypotension after adequate volume resuscitation and require vasopressor drugs to maintain a Mean Atrial Pressure (MAP) ≥ 65 mmHg and a serum lactate level > 2 mmol/L, it is considered that the sepsis patient has progressed to septic shock.

IPD SHARING:
Plan to Share IPD: No